CLINICAL TRIAL: NCT01149746
Title: A Single-Dose, Comparative Bioavailability Study of Two Formulations of Tamsulosin Hydrochloride 0.4 mg Capsules Under Fasting Conditions
Brief Title: Tamsulosin Hydrochloride 0.4 mg Capsules Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Responsible Party: Associate Director, Biopharmaceutics, Teva Pharmaceuticals USA
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2004-824
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tamsulosin (Experimental): 0.4 mg Capsule
  Interventions: Drug: Tamsulosin
- Flomax® (Active Comparator): 0.4 mg Capsule
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin — Test 0.4 mg Capsule
  Arms: Tamsulosin
Drug: Tamsulosin — Reference Listed 0.4 mg Capsule
  Other Names: Flomax®
  Arms: Flomax®

SUMMARY:
The objective of this study is to evaluate the comparative bioavailability between Tamsulosin Hydrochloride 0.4 mg Capsules (Teva Pharmaceuticals USA) and Flomax® 0.4 mg Capsules (Boehringer Ingelheim Pharmaceuticals, Inc. USA), after a single-dose in healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male subjects, 18 years of age or older.
* BMI greater than or equal to 19 and less than or equal to 30.
* Negative for:

  * HIV.
  * Hepatitis B surface antigen and Hepatitis C antibody.
  * Using drugs of abuse test (marijuana, amphetamines, barbiturates, cocaine, opiates, benzodiazepines and methadone).
  * Urine cotinine test
* No significant diseases or clinically significant findings in a physical examination.
* No clinically significant abnormal laboratory values.
* No clinically significant findings in vital signs measurements and a 12-lead electrocardiogram (ECG).
* Systolic blood pressure between 100-140 mmHg and diastolic blood pressure between 60-90 mmgHg.
* Be informed of the nature of the study and given written consent prior to receiving any study procedure.

Exclusion Criteria:

* Known history or presence of any clinically significant medical condition, illness or surgery within 4 weeks prior to drug administration.
* Known or suspected carcinoma.
* Known history or presence of:

  * Hypersensitivity or idiosyncratic reaction to tamsulosin and/or any other drug substances with similar activity.
  * Alcoholism within the last 12 months.
  * Drug dependence and/or substance abuse.
  * Use of tobacco or nicotine-containing products within the last 6 months.
* Use of any prescription medication within 14 days prior to Period 1 dosing. Use of any over the counter (OTC) medication within 7 days prior to Period 1 dosing.
* Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to Period 1 dosing.
* On a special diet within 4 weeks prior to drug administration (e.g. liquid, protein, raw food diet).
* Participated in another clinical trial or received and investigational product within 30 days prior to drug administration.
* Donated up to 250 mL of blood within the previous 30 days OR Donated from 251 to 500 mL of blood in the previous 45 days OR Donated more than 500 mL of blood in the previous 56 days (based on the Canadian Blood Services guideline for blood donation.
* Difficulty fasting or consuming the standard meals.
* Do not tolerate venipuncture.
* Unable to read or sign the ICF.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-12; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum observed concentration of drug substance in plasma) | Blood samples drawn over 60 hour time period
  Bioequivalence based on Cmax
AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration) | Blood samples drawn over 60 hour time period
  Bioequivalence based on AUC0-t
AUC0-inf (area under the concentration-time curve from time zero to infinity) | Blood samples drawn over 60 hour time period
  Bioequivalence based on AUC0-inf

CONTACTS AND LOCATIONS:
Overall Officials: Xueyu (Eric) Chen, M.D., Ph. D., FRCP (C), Principal Investigator — Pharma Medica Research, Inc.
Locations (1):
- Pharma Medica Research Inc., Toronto, Ontario, Canada